CLINICAL TRIAL: NCT04869904
Title: Analysis of the Periodontal Microbiota in Elderly Subjects With and Without Alzheimer's Disease: a Case Control Study
Brief Title: Oral Bacterial and Viral Mapping by Dental Plaque in Elderly Patients With and Without Alzheimer's Disease(ORal MICrobiology in Alzheimer's Patients)
Acronym: ORAMICAL
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 21Odonto02
Record Dates: First submitted 2021-04-27; First posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Periodontitis; Alzheimer Disease
MeSH Terms: conditions — Periodontitis; Alzheimer Disease | interventions — Dental Health Services

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva and plaque
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Alzheimer's disease
  Interventions: Procedure: dental and plaque sampling
- patients without Alzheimer's disease
  Interventions: Procedure: dental and plaque sampling

INTERVENTIONS:
Procedure: dental and plaque sampling — sampling of dental plaque and saliva during the treatment

SUMMARY:
The neurological disorders that accompany aging represent a major public health problem. The management of these diseases is a major medical and social priority. This project is based on the assumption that the oral cavity represents a privileged observation space to address these issues. The mouth is a site of easy access for painless sampling; there is therefore a major interest in identifying early oral infectious markers of the development or evolution of senile dementia. In addition to the interest of an early oral diagnosis, the mapping of the oral microbial flora in the demented elderly would allow a better understanding, prevention or even control of the evolution of neurodegenerative diseases. The final objective of our approach is to characterize the oral pathogens, or more probably the group of oral pathogens, which are significantly associated with Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 70 years old
* Patient (or trusted person) having read and understood the study information note and signed the informed consent form
* Membership in a social security scheme
* For cases : Diagnosis of possible or probable Alzheimer's disease according to the DSM-V

Exclusion Criteria:

* Presence of a neurodegenerative pathology (excluding Alzheimer's disease for cases)
* Presence of a neurocognitive disorder (excluding Alzheimer's disease for the cases)
* Patient with or having had any kind of cancer, including oral or aerodigestive tract
* Patients with or having had autoimmune diseases (HIV, hepatitis)
* Patients with inflammatory diseases (such as rheumatoid arthritis (RA) or Gougerot-Sjogren's syndrome (GSJ))
* Patients with severe haemopathy
* Patients with severe acute or chronic cardiovascular, renal, hepatic, gastrointestinal, allergic, endocrine, pulmonary, neuropsychiatric pathologies, judged by the investigator to be incompatible with the study, as all these pathologies may interfere with the results of the oral flora sampling
* Patients who have undergone oral surgery in the two months prior to sampling
* Patients treated with oral retinoids, bisphosphonates, oral anticoagulants or anticonvulsants
* Patients who have had anti-cancer or immunosuppressive chemotherapy within the last 6 months
* Patient who has had antibiotic or anti-inflammatory treatment in the last 4 weeks
* A history of treatments (drugs and probiotics) taken in the month prior to sampling will be taken, as well as a record of toxic habits (tobacco, alcohol, other)

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients coming to the Nice University Hospital (Autonomy Rehabilitation and Ageing Unit) for a memory consultation or a frailty screening
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Quantification of periodontal bacterial and viral species from dental plaque samples | 9 months
  Quantification of periodontal bacterial and viral species by microfluidic multiplex PCR-Biomark HD system Microfluidigm 9 Herpes viruses = HSV-1 and 2 (or HHV-1 and -2), VZV (or HHV-3), EBV (or HHV-4), CMV (or HHV-5), HHV-6A, HHV-6B, HHV-7, HHV-8 (or Kaposi virus) 16 periodontal bacteria = Porphyromonas gingivalis, Tannerella forsythensis, Treponema denticola, Prevotella intermedia, Campylobacter rectus, Fusobacterium nucleatum, Prevotella nigrescens, Eubacterium nodatum, Peptostreptococcus micros, Prevotella melaninogenica, Aa, Actinomyces naeslundii, Eikenella corrodens, Streptococcus mitis, Streptococcus oralis, Streptococcus sanguis
  For each species:
  Less than 25 CT (Cycle Treshold): positive More than 30 CT (Cycle Treshold): negative Between 25 and 30 CT (Cycle Treshold): need to increase significance by using an additional primer CT: allows to determine the number of copies of each bacterial or viral species

SECONDARY OUTCOMES:
Oral status presence of dentures | 9 Months
  presence of dentures: Yes/No masticatory coefficient: Coefficient from 1 to 5% assigned to each tooth according to its function, sum of all coefficients gives the result mobilities: Mühlemann index (from 0 to 3) caries involvement: DMFT
Oral status presence of dentures | 9 Months
  presence of dentures: Yes/No
Oral status masticatory coefficient | 9 Months
  presence of dentures: Yes/No masticatory coefficient: Coefficient from 1 to 5% assigned to each tooth according to its function, sum of all coefficients gives the result
Oral status mobilities | 1 day
  Mühlemann index (from 0 to 3)
Oral status caries involvement | 1 day
  DMFT: number of Decayed Missing or Filled teeth (from 0 to 32)
Periodontal status: pocket depth (PPS) | 9 months
  pocket depth (PPS): between the gum line and the bottom of the pocket, measures in mm.
Periodontal status: clinical attachment (CAL) | 9 months
  clinical attachment (CAL): between the enamel-cement junction and the bottom of the pocket, measures in mm.
Periodontal status: bleeding on probing (BOP): | 9 months
  bleeding on probing (BOP): number of sites with bleeding divided by total number of sites measured x 100, measured as a percentage.
Periodontal status: plaque index (PI) | 9 months
  plaque index (PI): from 0 to 3

CONTACTS AND LOCATIONS:
Locations (1):
- Nice University Hospital, Nice, France

IPD SHARING:
Plan to Share IPD: No